CLINICAL TRIAL: NCT01832584
Title: A Double-blind, Randomized, Placebo Controlled Study of the Effect of Red Grape Cells (RGC) Powder Consumption on Measures of Aerobic Fitness, Body Composition and Mood
Brief Title: Effect of Red Grape Cells (RGC) Powder Consumption on Measures of Aerobic Fitness and Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fruitura Bioscience Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: RGC-04
Record Dates: First submitted 2013-04-11; First posted 2013-04-16 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: Red Grapes; polyphenols; cyclists; resveratrol; aerobic fitness; trained

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- RGC1 (Experimental): 200 mg of Red Grape Cell (RGC) powder; daily oral dose
  Interventions: Dietary Supplement: RGC
- RGC2 (Experimental): 1000 mg of Red Grape Cell (RGC) powder; daily oral dose
  Interventions: Dietary Supplement: RGC
- Placebo (Placebo Comparator): 1000 mg placebo to Red Grape Cell (RGC) powder; daily oral dose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: RGC
  Other Names: Red Grape Cell powder
  Arms: RGC1; RGC2
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
This is a 3-arm double blind placebo controlled study to investigate the effect of Red Grape Cell (RGC) powder containing all the matrix of polyphenols that can be found in red grapes. polyphenols have several beneficial effects on various body systems, are present in many edible foods, and are considered safe for human consumption by regulatory authorities. Animal and human studies suggest a potential for polyphenol-rich compounds in enhancing mitochondrial activity and exercise capacity. However, the effect of RGC on exercise performance in humans had not yet been tested. A special population where increasing performance is highly sought are competitive athletes. The aim of the current study is to investigate the effect of RGC on measures of aerobic fitness, body composition and mood in trained male cyclists

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 65 years, men only
* Active in cycling training group
* Willingness to avoid regular use of NSAIDS (Advil, Nurofen, etc.) and aspirin for the entire study period
* Without a history or evidence of significant cardiovascular, hepatic, renal, respiratory, hematopoietic, gastrointestinal disease, endocrine, metabolic, psychiatric or psychological disorders;
* Willingness to avoid regular ingestion of any foods containing peanuts, bilberries, blueberries, cranberries, strawberries, raspberries, grapes, grape juice, cocoa powder, dark chocolate, red wine, over-the-counter medications, herbs, or supplements throughout the entire study, and to record and report any occasional consumption of such substances

Exclusion Criteria:

* Any acute medical situation (e.g., acute infection, nausea and vomiting, diarrhea) 48 hours prior to initiation of the study, which is considered of significance by the principal investigator.
* Any known chronic medical condition (will be determined by the principal investigator)
* History or evidence of alcohol or drug abuse
* Any gastrointestinal surgery other than appendectomy or herniotomy;
* Current use of over the counter or prescription weight loss medication
* Current use or within the last 30 days, any cholesterol lowering medications (statins, fibrates, red yeast rice, niacin).
* Known allergy to casein and/or soy.
* Subjects who had participated in a drug trial 3 months before initiation of the study;
* Non-cooperative subjects or unwilling to sign an informed consent and participate in the study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
changes in aerobic fitness | baseline and 6 weeks

SECONDARY OUTCOMES:
Changes in Body Mass Index (BMI) | baseline and 6 weeks
Changes in mood | baseline and 6 weeks
Changes in body weight | baseline and 6 weeks
Changes in body composition | baseline and 6 weeks
  changes in body fat percentage

OTHER OUTCOMES:
Number of adverse events | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gal Dubnov-Raz, M.D, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel